CLINICAL TRIAL: NCT05736068
Title: Is Casting of Displaced Pediatric Distal Forearm Fractures Non-inferior to Reduction in General Anesthesia? A Pragmatic, Randomized, Controlled Non-inferiority Multicenter Trial
Brief Title: Is Casting of Displaced Pediatric Distal Forearm Fractures Non-inferior to Reduction in General Anesthesia?
Acronym: CASTING
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Katrine Rønn Abildgaard, MD, PhD student, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-099-2022
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Distal Forearm Fracture; Distal Radius Fracture
Keywords: Forearm injuries; Wrist injuries; Salter-Harris fractures; Closed fracture reduction; Child; Bone remodeling
MeSH Terms: conditions — Wrist Fractures; Forearm Injuries; Wrist Injuries; Salter-Harris Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patient-Reported Outcome Measure (PROM) scores and radiographs will be evaluated by persons, who are blinded to treatment allocation and who are not otherwise involved in the study. Data analysis will be performed by an external biostatistician blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical (Experimental): No reduction. Application of a cast.
  Interventions: Procedure: Non-surgical treatment
- Surgical (Active Comparator): Closed reduction under general anesthesia with or without additional pin fixation of surgeons' choice followed by cast immobilization.
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Non-surgical treatment — If allocated to non-surgical group, cast optimization in the outpatient clinic may be necessary if the cast from the emergency room is considered insufficient.
  Arms: Non-surgical
Procedure: Surgical treatment — Closed reduction with or without fixation
  Arms: Surgical

SUMMARY:
Treatment of displaced distal forearm fractures (DFF) in children have traditionally been closed reduction and pin fixation, although they might heal and remodel without manipulation, with no functional impairment. No randomized controlled trials (RCTs) have been published comparing the patient-reported functional outcome after non-surgical and surgical treatment of displaced DFF in children.

This is a multicentre RCT. The aim of the trial is to investigate the patient-reported functional outcome after non-surgical treatment of displaced distal forearm fractures (DFF) in children. We will include 44 children aged 4-10 years with a displaced DFF. They will be offered inclusion, if the on-duty orthopedic surgeon finds indication for surgical intervention. If the parents/guardians consent to participate, the children will be allocated equally to non-surgical treatment (intervention) or surgical treatment of surgeon's choice (comparator). We will follow the children during one year, where they will be seen after 4 weeks, 3, 6 and 12 months. The primary outcome is the between-group difference in 12 months Quick Disabilities Arm Shoulder and Hand (QuickDASH) score.

DETAILED DESCRIPTION:
Pediatric distal forearm fractures (DFF) are very common and accounts for 25-30% of all fractures in children.(1,2) Up to half of all pediatric DFF are displaced to an extent where surgery has been the preferred treatment option.(3) However, surgery does come with a cost.

The most common treatment of displaced pediatric DFF has long been closed reduction with or without pin fixation (or in rare cases plate and screw fixation) under general anesthesia, followed by immobilization in a cast.(4) Pin-related complications vary from 4-23%, depending on what is reported as complications,(5-11) and up to 40% has been reported when including re-displacements.(12) The insertion of a metal wire or plate also requires subsequent procedures to remove these implants again.

Numerous small cohort studies and case series have found pin fixation advantageous in achieving anatomic reduction and avoiding re-displacement.(5-11) However, whether anatomic reduction and stabilization is important regarding the patient-reported functional outcome has not been investigated since most studies use only radiographic or objective measures (e.g. range of motion). In addition, children's bones, and in particular the metaphysis and epiphysis, have a unique ability to heal and remodel throughout the growth period until puberty.(13) Almost 20 years ago, Do et al. (14) stated that "the tremendous capacity of distal metaphyseal radius fractures to heal and remodel makes this one of the most rewarding fractures to treat non-operatively. […]". In accordance with Do et al., other studies indicate that displaced DFF fractures in prepubertal children might heal without manipulation, and that most displaced fractures will remodel within a year or two to almost anatomical position with no functional impairment.(14-17) Although most surgeons are aware that children's bones have this remodeling potential, they still find it challenging to deal with the uncertainty of whether the bone will actually remodel to an acceptable position. Furthermore, surgeons might have difficulties with how families will react to the waiting time until the misaligned arm looks normal again.

If non-surgical treatment of displaced pediatric DFF were more common, the costs associated with surgery could be minimized. Unfortunately, there is limited evidence to guide the decision to operate or not. The available studies are typically small, retrospective cohort studies or case series of low quality with no predefined follow-up or outcome measures. To our knowledge, there are no published randomized controlled trials (RCTs) comparing non-surgical treatment with surgical treatment, and no studies report outcomes from the patient's perspective.

The aim of this trial is to investigate the patient-reported functional outcome after non-surgical treatment of displaced DFF in children aged 4-10 years. Our hypothesis is, that casting without manipulation is non-inferior to surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-10 years of age with open physes
* Fractures in the distal metaphyseal radius (with or without concomitant ulna fracture), including extraarticular physeal fractures (SH I-II)

  * Overriding fractures
  * Angulated fractures of 20-40°
* The on-duty surgeon finds reduction under anesthesia with or without fixation indicated

Exclusion Criteria:

* Open fractures
* Nerve or vascular affection
* All intraarticular fractures including SH III-V
* Ulnar physeal fractures
* Polytrauma
* Concomitant ipsi- or contralateral upper extremity fractures (except distal ulna fracture)
* Pathologic fractures
* The injury is >7 days old
* Other conditions that may affect bone healing

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
QuickDASH | 12 months
  Reporting of disability experienced and monitoring changes in symptoms and function over time. The patient (with help by parents if the patient is too young to self-report) rates each item according to the perceived degree of severity using a 5-point Likert Scale. Then, the overall score is transformed to a score between 0 and 100 (0 = no disability, 100 = maximum disability) according to the algorithm [(sum of responses N/N)-1]*25, where N is equal to the number of responses.

SECONDARY OUTCOMES:
QuickDASH | 3 and 6 months
  Reporting of disability experienced and monitoring changes in symptoms and function over time. The patient (with help by parents if the patient is too young to self-report) rates each item according to the perceived degree of severity using a 5-point Likert Scale. Then, the overall score is transformed to a score between 0 and 100 (0 = no disability, 100 = maximum disability) according to the algorithm [(sum of responses N/N)-1]*25, where N is equal to the number of responses.
EQ-5D-Y | 3, 6 and 12 months
  Health-related quality of life. The questionnaire consists of two parts:
  1. the descriptive system which assesses health in five dimensions (Mobility; Looking After Myself; Doing Usual Activities; Having Pain or Discomfort; Feeling Worried, Sad or Unhappy).
  2. A visual analogue scale (VAS) on which the respondent rates their perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health)
Wong-Baker Faces Pain Rating Scale (WBS) | 3, 6 and 12 months
  A self-reported tool to assess pain using a series of six facial expressions to illustrate the degree of pain intensity.

OTHER OUTCOMES:
Radiographs (explorative outcome) | 6 and 12 months
  Evaluation of the remodeling process. No statistical analysis will be made.
Photographs (explorative outcome) | 3, 6 and 12 months
  Observation of the cosmetic progress and to be used for documentation of what future patients can expect cosmetically.

CONTACTS AND LOCATIONS:
Overall Officials: Stig Brorson, MD PhD DMSc, Study Director — Zealand University Hospital; Katrine R. Abildgaard, MD, Principal Investigator — Zealand University Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Zealand University Hospital, Køge
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedstrom EM, Svensson O, Bergstrom U, Michno P. Epidemiology of fractures in children and adolescents. Acta Orthop. 2010 Feb;81(1):148-53. doi: 10.3109/17453671003628780. PMID 20175744
- [Background] Hove LM, Brudvik C. Displaced paediatric fractures of the distal radius. Arch Orthop Trauma Surg. 2008 Jan;128(1):55-60. doi: 10.1007/s00402-007-0473-x. Epub 2007 Oct 17. PMID 17940779
- [Background] Laaksonen T, Kosola J, Nietosvaara N, Puhakka J, Nietosvaara Y, Stenroos A. Epidemiology, Treatment, and Treatment Quality of Overriding Distal Metaphyseal Radial Fractures in Children and Adolescents. J Bone Joint Surg Am. 2022 Feb 2;104(3):207-214. doi: 10.2106/JBJS.21.00850. PMID 34780389
- [Background] Handoll HH, Elliott J, Iheozor-Ejiofor Z, Hunter J, Karantana A. Interventions for treating wrist fractures in children. Cochrane Database Syst Rev. 2018 Dec 19;12(12):CD012470. doi: 10.1002/14651858.CD012470.pub2. PMID 30566764
- [Background] Proctor MT, Moore DJ, Paterson JM. Redisplacement after manipulation of distal radial fractures in children. J Bone Joint Surg Br. 1993 May;75(3):453-4. doi: 10.1302/0301-620X.75B3.8496221.
- [Background] McLauchlan GJ, Cowan B, Annan IH, Robb JE. Management of completely displaced metaphyseal fractures of the distal radius in children. A prospective, randomised controlled trial. J Bone Joint Surg Br. 2002 Apr;84(3):413-7. doi: 10.1302/0301-620x.84b3.11432. PMID 12002503
- [Background] Gibbons CL, Woods DA, Pailthorpe C, Carr AJ, Worlock P. The management of isolated distal radius fractures in children. J Pediatr Orthop. 1994 Mar-Apr;14(2):207-10. doi: 10.1097/01241398-199403000-00014. PMID 8188835
- [Background] Wendling-Keim DS, Wieser B, Dietz HG. Closed reduction and immobilization of displaced distal radial fractures. Method of choice for the treatment of children? Eur J Trauma Emerg Surg. 2015 Aug;41(4):421-8. doi: 10.1007/s00068-014-0483-7. Epub 2014 Dec 19. PMID 26038007
- [Background] Colaris JW, Allema JH, Biter LU, de Vries MR, van de Ven CP, Bloem RM, Kerver AJ, Reijman M, Verhaar JA. Re-displacement of stable distal both-bone forearm fractures in children: a randomised controlled multicentre trial. Injury. 2013 Apr;44(4):498-503. doi: 10.1016/j.injury.2012.11.001. Epub 2012 Dec 3. PMID 23217981
- [Background] Zamzam MM, Khoshhal KI. Displaced fracture of the distal radius in children: factors responsible for redisplacement after closed reduction. J Bone Joint Surg Br. 2005 Jun;87(6):841-3. doi: 10.1302/0301-620X.87B6.15648. PMID 15911670
- [Background] McQuinn AG, Jaarsma RL. Risk factors for redisplacement of pediatric distal forearm and distal radius fractures. J Pediatr Orthop. 2012 Oct-Nov;32(7):687-92. doi: 10.1097/BPO.0b013e31824b7525. PMID 22955532
- [Background] Miller BS, Taylor B, Widmann RF, Bae DS, Snyder BD, Waters PM. Cast immobilization versus percutaneous pin fixation of displaced distal radius fractures in children: a prospective, randomized study. J Pediatr Orthop. 2005 Jul-Aug;25(4):490-4. doi: 10.1097/01.bpo.0000158780.52849.39. PMID 15958902
- [Background] Wilkins KE. Principles of fracture remodeling in children. Injury. 2005 Feb;36 Suppl 1:A3-11. doi: 10.1016/j.injury.2004.12.007. PMID 15652934
- [Background] Do TT, Strub WM, Foad SL, Mehlman CT, Crawford AH. Reduction versus remodeling in pediatric distal forearm fractures: a preliminary cost analysis. J Pediatr Orthop B. 2003 Mar;12(2):109-15. doi: 10.1097/01.bpb.0000043725.21564.7b. PMID 12584495
- [Background] Laaksonen T, Puhakka J, Stenroos A, Kosola J, Ahonen M, Nietosvaara Y. Cast immobilization in bayonet position versus reduction and pin fixation of overriding distal metaphyseal radius fractures in children under ten years of age: a case control study. J Child Orthop. 2021 Feb 1;15(1):63-69. doi: 10.1302/1863-2548.15.200171. PMID 33643460
- [Background] Marson BA, Ng JWG, Craxford S, Chell J, Lawniczak D, Price KR, Ollivere BJ, Hunter JB. Treatment of completely displaced distal radial fractures with a straight plaster or manipulation under anaesthesia. Bone Joint J. 2021 May;103-B(5):902-907. doi: 10.1302/0301-620X.103B.BJJ-2020-1740.R1. Epub 2021 Mar 12. PMID 33709769
- [Background] Crawford SN, Lee LS, Izuka BH. Closed treatment of overriding distal radial fractures without reduction in children. J Bone Joint Surg Am. 2012 Feb 1;94(3):246-52. doi: 10.2106/JBJS.K.00163. PMID 22298057
- [Background] Meling T, Harboe K, Enoksen CH, Aarflot M, Arthursson AJ, Soreide K. Reliable classification of children's fractures according to the comprehensive classification of long bone fractures by Muller. Acta Orthop. 2013 Apr;84(2):207-12. doi: 10.3109/17453674.2012.752692. Epub 2012 Dec 18. PMID 23245225
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Gummesson C, Ward MM, Atroshi I. The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): validity and reliability based on responses within the full-length DASH. BMC Musculoskelet Disord. 2006 May 18;7:44. doi: 10.1186/1471-2474-7-44. PMID 16709254
- [Background] Quatman-Yates CC, Gupta R, Paterno MV, Schmitt LC, Quatman CE, Ittenbach RF. Internal consistency and validity of the QuickDASH instrument for upper extremity injuries in older children. J Pediatr Orthop. 2013 Dec;33(8):838-42. doi: 10.1097/BPO.0b013e3182a00688. PMID 23863415
- [Background] Gao B, Dwivedi S, Patel SA, Nwizu C, Cruz AI Jr. Operative Versus Nonoperative Management of Displaced Midshaft Clavicle Fractures in Pediatric and Adolescent Patients: A Systematic Review and Meta-Analysis. J Orthop Trauma. 2019 Nov;33(11):e439-e446. doi: 10.1097/BOT.0000000000001580. PMID 31633645
- [Background] Roper B, Parikh S, Haidar L, Warth R, Ambrose C, Younas S, Crawford L, Mansour A. Outcomes After Operative Treatment of Pediatric Monteggia Fracture-Dislocations: Comparison Between Open and Closed Injuries. J Pediatr Orthop. 2022 Aug 1;42(7):361-366. doi: 10.1097/BPO.0000000000002171. Epub 2022 May 10. PMID 35543603
- [Background] Eguia F, Gottlich C, Lobaton G, Vora M, Sponseller PD, Lee RJ. Mid-term Patient-reported Outcomes After Lateral Versus Crossed Pinning of Pediatric Supracondylar Humerus Fractures. J Pediatr Orthop. 2020 Aug;40(7):323-328. doi: 10.1097/BPO.0000000000001558. PMID 32271317
- [Background] Ernat J, Ho C, Wimberly RL, Jo C, Riccio AI. Fracture Classification Does Not Predict Functional Outcomes in Supracondylar Humerus Fractures: A Prospective Study. J Pediatr Orthop. 2017 Jun;37(4):e233-e237. doi: 10.1097/BPO.0000000000000889. PMID 27776052
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Sorensen AA, Howard D, Tan WH, Ketchersid J, Calfee RP. Minimal clinically important differences of 3 patient-rated outcomes instruments. J Hand Surg Am. 2013 Apr;38(4):641-9. doi: 10.1016/j.jhsa.2012.12.032. Epub 2013 Mar 6. PMID 23481405
- [Background] Polson K, Reid D, McNair PJ, Larmer P. Responsiveness, minimal importance difference and minimal detectable change scores of the shortened disability arm shoulder hand (QuickDASH) questionnaire. Man Ther. 2010 Aug;15(4):404-7. doi: 10.1016/j.math.2010.03.008. PMID 20434942
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Background] Wille N, Badia X, Bonsel G, Burstrom K, Cavrini G, Devlin N, Egmar AC, Greiner W, Gusi N, Herdman M, Jelsma J, Kind P, Scalone L, Ravens-Sieberer U. Development of the EQ-5D-Y: a child-friendly version of the EQ-5D. Qual Life Res. 2010 Aug;19(6):875-86. doi: 10.1007/s11136-010-9648-y. Epub 2010 Apr 20. PMID 20405245
- [Background] Ravens-Sieberer U, Wille N, Badia X, Bonsel G, Burstrom K, Cavrini G, Devlin N, Egmar AC, Gusi N, Herdman M, Jelsma J, Kind P, Olivares PR, Scalone L, Greiner W. Feasibility, reliability, and validity of the EQ-5D-Y: results from a multinational study. Qual Life Res. 2010 Aug;19(6):887-97. doi: 10.1007/s11136-010-9649-x. Epub 2010 Apr 17. PMID 20401552
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Verstraete J, Lloyd A, Scott D, Jelsma J. How does the EQ-5D-Y Proxy version 1 perform in 3, 4 and 5-year-old children? Health Qual Life Outcomes. 2020 May 24;18(1):149. doi: 10.1186/s12955-020-01410-3. PMID 32448278
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Phelps EE, Tutton E, Costa ML, Achten J, Moscrop A, Perry DC. Protecting my injured child: a qualitative study of parents' experience of caring for a child with a displaced distal radius fracture. BMC Pediatr. 2022 May 12;22(1):270. doi: 10.1186/s12887-022-03340-z. PMID 35549910
- [Derived] Abildgaard KR, Buxbom P, Rahbek O, Gottliebsen M, Gundtoft PH, Viberg B, Brorson S. Is casting of displaced paediatric distal forearm fractures non-inferior to reduction under general anaesthesia? Study protocol for a pragmatic, randomized, controlled non-inferiority multicentre trial (the casting trial). Trials. 2024 Jun 27;25(1):420. doi: 10.1186/s13063-024-08253-z. PMID 38937792